CLINICAL TRIAL: NCT05657353
Title: Correlation Between Bruxism And Cervical Function
Brief Title: Relation Between Bruxism and Cervical Function
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Olivia Ibrahim Abdelmesseh Angly, Doctor of physical therapy, Cairo University
Other Study IDs: Bruxism And Cervical Function
Record Dates: First submitted 2022-11-28; First posted 2022-12-20 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Bruxism
Keywords: Bruxism; cervical pain; cervical proprioception
MeSH Terms: conditions — Bruxism; Neck Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
correlation between Bruxism and Cervical function

DETAILED DESCRIPTION:
Bruxism is defined as an unconscious oral habit of dysfunctional rhythmic pressing, clenching and grinding of the teeth when performing movements that are not part of the masticatory function that leads to occlusal trauma and it is an oral parafunctional activity it is not related to normal physiological functions, such as speech, breathing, chewing and swallowing , and/or by bracing or thrusting of the mandible , and it accelerates abnormal tooth wear, periodontal disease, and temporomandibular disorders (TMD)

Bruxism should be considered a potential protective risk factor rather than a disorder in otherwise healthy individuals. In most persons bruxism is not a disorder, it is a sign of a disorder (e.g. in individuals with obstructive sleep apnea, epilepsy , being the ending episode of respiratory arousals, so as to prevent the collapse or restore the patency of the upper airway whilst asleep) , which would classify bruxism as an attribute that decreases the chance of a negative health outcome.

There is two distinct circadian manifestations, either occurring during wakefulness or during sleep. Awake bruxism is a semivoluntary masticatory muscle activity during wakefulness that is characterized clenching or grinding tooth and/or by bracing or thrusting of the mandible

ELIGIBILITY:
Inclusion Criteria:

* Tooth-grinding or clenching .
* Sounds associated with bruxism or jaw muscle discomfort.
* Pain in the jaw, temple, ear or front of the ear and pain modified by jaw movement, function, or parafunction.

Exclusion Criteria:

* History of trauma to the face .
* History of orthodontic treatment, craniofacial anomalies, degenerative disease, or TMJ trauma .
* Any systematic joint or muscle disease and neurologic disorder. neurologic disorders (eg, trigeminal neuralgi ,neurologic disorders (eg, trigeminal neuralgi neurologic disorders (eg, trigeminal neuralgi
* Osteoarthrosis or arthritis of temporomandibular joint .
* Tumors in the head and neck area.

Ages: 18 Years to 30 Years | Sex: All
Age Groups: Adult
Study Population: Observational Cohort Study
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Pressure Algometer | 4 months
  to measure pain threshold of masseter and temporalis and sternocledomastoid trigger points

SECONDARY OUTCOMES:
Bubble Incliniometer | 4 months
  to measure cervical proprioception in flexion ,extension and right and left rotation

CONTACTS AND LOCATIONS:
Overall Officials: Rania karkousha, Assis.Prof., Principal Investigator — university
Locations (1):
- IPC clinic, Giza, Egypt